CLINICAL TRIAL: NCT05604443
Title: Keratoconus Detection Using MS39 and Pentacam - a Retrospective Study
Brief Title: Keratoconus Detection Using MS39 and Pentacam
Acronym: KKMS39Penta
Status: Completed | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: KUK-Ophthalmology-007
Record Dates: First submitted 2022-10-05; First posted 2022-11-03 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Keratoconus
Keywords: Keratoconus; Pentacam; MS39
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective analyze — retrospective analyze of MS39 and Pentacam images

SUMMARY:
This retrospective study aims to investigate whether the MS39 and Pentacam are delivering comparable results in the diagnosis of keratoconus.

In the future, these measurement devices could be interchangeable in usage.

DETAILED DESCRIPTION:
Keratoconus is a degenerative pathology of the cornea, which tends to progress. It comes along with central and paracentral thinning of the cornea as well as with an apical protrusion of the cornea. Keratoconus leads to vision loss. This pathology is diagnosed by using CE certified OCT technology in order to map the topography of the cornea. This process constitutes a really important step in the line of management of the keratoconus. MS39 and Pentacam are used for detection. Retrospectively, data will be investigated, in order to see if these measurement devices deliver comparable results. In the future, these measurement devices could be interchangeable in usage.

ELIGIBILITY:
Inclusion Criteria:

* age older than 14 years
* patients who show up at Keratokonus consultation hours

Exclusion Criteria:

* age younger than 14 years
* age older than 100 years

Ages: 14 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients between 14 and 100 years who consult Keratokonus specialst.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
topography of the cornea | 12 months
  measurement of the topography of the cornea with MS39 and Pentacam

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bolz, MD, Principal Investigator — JKU Linz
Locations (1):
- Department for Ophthalmology and Optometry, Kepler University Hospital GmbH, Johannes Kepler University Linz, Altenberger Strasse 69, 4040 Linz, Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No